CLINICAL TRIAL: NCT01876303
Title: Genetic Epidemiology of Ewing's Sarcoma
Brief Title: Genetic Biomarkers in Saliva Samples From Patients With Ewing Sarcoma
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AEPI10N5; NCI-2012-02210 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); AEPI10N5 (Other: Children's Oncology Group); AEPI10N5 (Other: CTEP); U10CA098543 (NIH)
Record Dates: First submitted 2013-06-10; First posted 2013-06-12 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Ewing Sarcoma/Peripheral Primitive Neuroectodermal Tumor (PNET)
MeSH Terms: conditions — Neuroectodermal Tumors, Primitive, Peripheral

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — saliva
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ancillary-Correlative (genetic epidemiology of Ewing sarcoma): Genomic DNA is extracted from participants' saliva samples and analyzed for expression of EWS-FLI1 and other ES-target genes.
  Interventions: Other: laboratory biomarker analysis; Other: questionnaire administration

INTERVENTIONS:
Other: laboratory biomarker analysis — Correlative studies
Other: questionnaire administration — Ancillary studies

SUMMARY:
This clinical trial studies genetic biomarkers from saliva samples in patients with Ewing sarcoma. Studying samples of saliva from patients with cancer in the laboratory may help doctors learn more about changes that occur in deoxyribonucleic acid (DNA) and identify biomarkers related to cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the association between the length of Ewing sarcoma breakpoint region 1-Friend leukemia virus integration 1 (EWS-FLI1) fusion protein binding sites (microsatellites) and risk of Ewing's sarcoma (ES).

II. To determine the frequency and commonality of Caucasian ancestral markers in cases of ES self-identified as non-Caucasian (African-American, Asian, Hispanic).

III. To determine the association between genomic variants in ES-related genes and hernia development (i.e. the integrin signaling pathway) and risk of ES.

OUTLINE:

Genomic DNA is extracted from participants' saliva samples and analyzed for expression of EWS-FLI1 and other ES-target genes.

ELIGIBILITY:
Inclusion Criteria:

* The patient is enrolled on ACCRN07
* The patient has a diagnosis of Ewing Sarcoma (International Classification of Diseases [ICD] code morphology 9260; topography C40.0-C41.9, C76.0-C76.8, C80.9) and is registered with Children's Oncology Group (COG) by a North American member institution
* The patient must be diagnosed with Ewing sarcoma between December 24, 2007 and December 31, 2015
* The patient must have at least one biological parent alive and willing to participate
* All questionnaire respondents must understand English or Spanish
* Concomitant treatment on a therapeutic trial is not required

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a diagnosis of Ewing Sarcoma meeting other criteria.
Sampling Method: Non-Probability Sample
Enrollment: 1650 (Estimated)
Dates: Start 2012-12; Primary Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Main effect of gene polymorphisms | Up to 5 years
  Risk ratios (RR) for the main effect of gene polymorphisms will be calculated using log-linear models. RRs and 95% confidence intervals for the gene-environment interaction are calculated by stratifying the likelihood according to case exposure.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Schiffman, MD, Principal Investigator — Children's Oncology Group
Locations (1):
- Children's Oncology Group, Monrovia, California, United States

REFERENCES:
- [Derived] Zieger HK, Weinhold L, Schmidt A, Holtgrewe M, Juranek SA, Siewert A, Scheer AB, Thieme F, Mangold E, Ishorst N, Brand FU, Welzenbach J, Beule D, Paeschke K, Krawitz PM, Ludwig KU. Prioritization of non-coding elements involved in non-syndromic cleft lip with/without cleft palate through genome-wide analysis of de novo mutations. HGG Adv. 2022 Dec 5;4(1):100166. doi: 10.1016/j.xhgg.2022.100166. eCollection 2023 Jan 12. PMID 36589413